CLINICAL TRIAL: NCT06757426
Title: Prospective Observational Study Evaluating the Safety and Efficacy of Immunomodulatory Therapies in Refractory Inflammatory and Autoimmune Diseases
Acronym: ARIES
Status: Not yet recruiting | Type: Observational
Sponsor: Groupe français d'étude des Maladies Inflammatoires de loeil (Other)
Responsible Party: Sponsor
Other Study IDs: ARIES; 2024-A02472-45 (Other: ANSM)
Record Dates: First submitted 2024-12-18; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Diseases; Inflammatory Diseases
Keywords: autoimmune; inflamatory disease; Refraction
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with immune-mediated inflammatory disease refractory to conventional lines of therapy: Adult patients with immune-mediated inflammatory disease refractory to conventional lines of therapy.

SUMMARY:
Inflammatory and/or autoimmune diseases represent a very broad group of diseases with highly variable clinical features, including - but not limited to - systemic connectivites and vasculitides. As these diseases are rare and heterogeneous, it is difficult to conduct randomized clinical trials in this setting. Refractory cases are therefore treated with drugs that are already available on the market for other indications in more frequent and clinically homogeneous diseases, such as inflammatory rheumatism and haematological malignancies.

Prescribing treatments from other specialties (e.g. rheumatology and oncohaematology) is a reality in the clinical practice of internists and immunologists, often representing an excellent solution for difficult-to-treat inflammatory and/or autoimmune diseases. As these molecules are prescribed without the availability of standardized data, it is essential to collect them prospectively to better characterize the efficacy and tolerability of these new therapeutic options in severe inflammatory and/or autoimmune diseases.

DETAILED DESCRIPTION:
Inflammatory and/or autoimmune diseases represent a very broad group of diseases with highly variable clinical features, including - but not limited to - systemic connectivites and vasculitis. Individually, they are very rare diseases, generally estimated in terms of the number of cases per 100,000 or 1,000,000 inhabitants. However, if we consider all immune-mediated inflammatory diseases, it is estimated that they affect 4.5% of the world's population .

Despite their extreme heterogeneity in terms of clinical presentation, these diseases share several key pathogenic mechanisms. For example, over the past two decades, adaptive immunity has been successfully targeted with several monoclonal antibodies directed against B lymphocytes (e.g. rituximab, an anti-CD20) and co-stimulation between B and T lymphocytes (e.g. abatacept, a CTLA-4 agonist). Targeting cytokines common to several of these diseases has also proved effective in their management, in particular anti-TNF alpha and anti-IL-6, produced by cells of the innate and adaptive immune systems.

Although these molecules have ushered in a new era in the management of inflammatory and/or autoimmune diseases, not all patients are yet fully controlled, representing a major challenge in clinical practice.

Refractory cases are then treated with drugs that are already available on the market for other indications in more frequent and clinically homogeneous diseases, such as inflammatory rheumatism and haematological malignancies.

Certain therapeutic targets stand out. The first is the cytokine IL-17, which plays a crucial role in the polarization of T helper 17 (Th17) lymphocytes and orchestrates the adaptive response detectable in the blood and target tissues of various inflammatory and/or autoimmune diseases.

Another interesting modern strategy is the inhibition of the Janus kinase and signal transducer/activator of transcription (JAK/STAT) pathways, which act on several downstream cytokine receptors. The development of targeted oral therapies based on small molecules such as JAK inhibitors (JAKi) represents an effective means of simultaneously attenuating several downstream inflammatory pathways, and has enabled a paradigm shift in the treatment of various autoimmune and inflammatory conditions refractory to conventional therapy, with cortisone sparing as well.

Bispecific antibodies (BsAb) are a new class of drugs and one of the most promising immunotherapies for solid tumors and hematological malignancies. BsAbs combine the specificities of two therapeutic antibodies and simultaneously target different antigens or epitopes. They have attracted a great deal of interest over the past decade, thanks to their unique and versatile modes of action.

In summary, the prescription of commercially available treatments from other specialties (e.g. rheumatology and oncohaematology) is a reality in the clinical practice of internists and immunologists, often representing an excellent solution for difficult-to-treat inflammatory and/or autoimmune diseases. As these molecules are prescribed without the availability of standardized data, it is essential to collect them prospectively to better characterize the efficacy and tolerability of these new therapeutic options in inflammatory and/or autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years
2. Enrolled in the French national social security system
3. Diagnosis of an inflammatory/autoimmune disease meeting internationally accepted classification criteria;
4. Clinical activity of their disease with biological and/or radiological signs, refractory to conventional therapeutic lines, requiring a new treatment as an addition or replacement according to clinical judgment.
5. No formal contraindication to the new therapeutic class.

Exclusion Criteria:

1. Pregnancy or breast-feeding (for women of childbearing potential, a negative serum pregnancy test will be required);
2. History of severe immunosuppression, HIV or HBsAg positive.
3. Positive QuantiFERON test result (QFT-TBGIn-Tube) for active tuberculosis (latent tuberculosis under treatment may be included).
4. Have received live vaccines in the 3 months preceding the start of treatment.
5. History of malignant tumor within the last 5 years.
6. Severe renal insufficiency (creatinine clearance <30mL/min/1.73m²)
7. Liver dysfunction defined by aspartate transaminase (AST) or alanine transaminase (ALT) levels ≥ 5 times the upper limit of normal.
8. Blood count abnormality:

   * Platelets < 50 x 103/mm3
   * Neutropenia < 1000/mm3
   * Hemoglobin < 8 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory inflammatory and autoimmune diseases
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
proportion of complete remission from the disease at week 24 | week 24
  The primary outcome will be the proportion of complete remission from the disease at week 24 :
  1. absence of all clinical signs and symptoms ;
  2. normalization of fibrinogen and CRP values;
  3. absence of radiological signs of active disease (stable or improved imaging).

SECONDARY OUTCOMES:
Evaluate the proportion of patients in clinical, biological or radiological remission | week 12 and week 48
  Evaluate the proportion of patients with clinical remission (endpoint #1 of the primary endpoint), biological remission (endpoint #2 of the primary endpoint) or radiological remission (endpoint #3 of the primary endpoint) at weeks 12 and 48 of the indicated treatment start.
Cumulative incidence of relapse (i.e., recurrence of clinical symptoms associated with biological and/or radiological inflammatory activity following complete remission) | weeks 12, 24, 36 and 52
  Cumulative incidence of relapse (i.e., recurrence of clinical symptoms associated with biological and/or radiological inflammatory activity following complete remission) at weeks 12, 24, 36 and 52;
Cumulative incidence of remission according to primary endpoint definitions | weeks 12, 36 and 52
  Cumulative incidence of remission according to primary endpoint definitions at weeks 12, 36 and 52
Evaluate changes in median disease-specific activity scores | weeks 12, 24, 36 and 52
  Evaluate changes in median disease-specific activity scores at weeks 12, 24, 36 and 52
Cumulative prednisone dose | weeks 12, 24, 36 and 52
  Cumulative prednisone dose at weeks 12, 24, 36 and 52
Cumulative incidence of serious adverse events (i.e., those requiring hospitalization or death) at weeks 12, 24, 36 and 52 | weeks 12, 24, 36 and 52
  Cumulative incidence of serious adverse events (i.e., those requiring hospitalization or death) at weeks 12, 24, 36 and 52
Evolution of circulating immune cell populations & cytokines under treatment | Weeks 0, 1, 2, 4, 12, 24, and 52
  Evolution of circulating immune cell populations & cytokines under treatment by measuring the change in the proportion of B & T cells & cytokines in peripheral blood before, during and following treatment.

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Clinique Axium - Aix-en-provence, Aix-en-Provence
  - CH Simone Veil de BLOIS, Blois
  - CHU Caen Normandie, Caen
  - CH du Mans, Le Mans
  - APHM_Hôpital La Conception, Marseille
  - APHM_Hôpital Nord, Marseille
  - GHSIF Melun, Melun
  - GHI Le Raincy Montfermeil, Montfermeil
  - CHU Nantes - Hotel-Dieu, Nantes
  - CHU Rouen_Hôpital Charles Nicolle, Rouen
  - Clinique Saint-Exupéry, Saint-Exupéry
  - CHRU de Tours_Hôpital Bretenneau, Tours
  - APHP_Hopital Lariboisière, Paris, Île-de-France Region
  - APHP_Hôpital St Antoine, Paris, Île-de-France Region
  - APHP_ Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region
  - APHP_Hôpital Bichat, Paris, Île-de-France Region
  - APHP_Hopital Ambroise Paré, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Venhoff N, Schmidt WA, Bergner R, Rech J, Unger L, Tony HP, Finzel S, Andreica I, Kofler DM, Weiner SM, Lamprecht P, Schulze-Koops H, App C, Pournara E, Mendelson MH, Sieder C, Maricos M, Thiel J. Safety and efficacy of secukinumab in patients with giant cell arteritis (TitAIN): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2023 Jun;5(6):e341-e350. doi: 10.1016/S2665-9913(23)00101-7. PMID 38251601
- [Background] Klein C, Brinkmann U, Reichert JM, Kontermann RE. The present and future of bispecific antibodies for cancer therapy. Nat Rev Drug Discov. 2024 Apr;23(4):301-319. doi: 10.1038/s41573-024-00896-6. Epub 2024 Mar 6. PMID 38448606
- [Background] Hayter SM, Cook MC. Updated assessment of the prevalence, spectrum and case definition of autoimmune disease. Autoimmun Rev. 2012 Aug;11(10):754-65. doi: 10.1016/j.autrev.2012.02.001. Epub 2012 Feb 23. PMID 22387972
- [Background] Watts RA, Hatemi G, Burns JC, Mohammad AJ. Global epidemiology of vasculitis. Nat Rev Rheumatol. 2022 Jan;18(1):22-34. doi: 10.1038/s41584-021-00718-8. Epub 2021 Dec 1. PMID 34853411
- See also: LBA0001 EFFICACY AND SAFETY OF UPADACITINIB IN PATIENTS WITH GIANT CELL ARTERITIS (SELECT-GCA): A DOUBLE-BLIND, RANDOMIZED CONTROLLED PHASE 3 TRIAL — https://ard.bmj.com/content/83/Suppl_1/232